CLINICAL TRIAL: NCT05393934
Title: Clinical Trial on Intervention Growth Faltering Using Pediatric Nutritional Care Compared to Pediatric Nutritional Care and Food for Special Medical Purposes (FSMP)
Brief Title: Growth Faltering Intervention Using Pediatric Nutritional Care (PNC) vs.PNC& FSMP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Specialized Nutrition Indonesia (Industry)
Collaborators: Hasanuddin University (Other); RIKEN (Other); LMU Klinikum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 010322
Record Dates: First submitted 2022-04-04; First posted 2022-05-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Growth Failure
MeSH Terms: conditions — Failure to Thrive | interventions — Food

STUDY DESIGN:
Intervention Model Description: Non randomized and controlled study design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PNC (Pediatric Nutrition Care) (Placebo Comparator): This first group will be given pediatric nutrition care (PNC) in visit 0. In this group parents will receive nutritional advice about how many calories are needed, the type and form of food that can be given so that the baby can gain weight accordingly.
  Interventions: Other: Pediatric Nutrition Care (PNC)
- FSMP (Food for Special Medical Purposes) & PNC (Pediatric Nutrition Care) (Active Comparator): In this second group, subject will receive PNC in visit 0 and food for special medically purposes/FSMP that will be given according to daily calorie needs which are determined based on ideal body weight (BB) according to body length. In general, FSMP will be given 3 times a day, according to the needs of each subject. Parents will be taught about preparation of FSMP e.g. dissolving and the correct amount of product (image will be attached in the appendix). FSMP will be given during the research period and will be discontinued when not needed anymore.
  Interventions: Other: High dense nutrients formula; Other: Pediatric Nutrition Care (PNC)

INTERVENTIONS:
Other: High dense nutrients formula — High dense nutrients formula: Powder based Infant formula with High Nutrients' Density with energy density of 100 kcal/100ml and for Pediatric Nutrition Care: A medical service to understand nutritional status, problems related to the feeding process and clinical diagnosis of the patient.
  Other Names: food for special medically purposes
  Arms: FSMP (Food for Special Medical Purposes) & PNC (Pediatric Nutrition Care)
Other: Pediatric Nutrition Care (PNC) — Pediatric Nutrition Care: A medical service to understand nutritional status, problems related to the feeding process and clinical diagnosis of the patient.

SUMMARY:
Study will be done by consortium of pediatrician from Indonesia, Japan, and Germany. This team will act as leaders while the field assistant will consist of nutritionist and general practitioner. The chosen primary endpoint is the improvement of weight for age (grams) of the sample after one month of intervention. Participants are weight faltering babies aged 6-12 months at study entry, with the weight increments below P 15th of WHO weight increments tables whose parents agreed to be included in the study by providing written informed consent.

DETAILED DESCRIPTION:
Study will be done by consortium of pediatrician from Indonesia, Japan, and Germany. This team will act as leaders while the field assistant will consist of nutritionist and general practitioner. The chosen primary endpoint is the improvement of weight for age (grams) of the sample after one month of intervention. Participants are weight faltering babies aged 6-12 months at study entry, with the weight increments below P 15th of WHO weight increments tables whose parents agreed to be included in the study by providing written informed consent. The investigators aim to include 2 x 94 babies for a randomized control trial study residing in Makassar, South Sulawesi. They will be selected and enrolled after matching for age and sex. All babies will be examined in for their nutritional status, demographics, medical history, preexisting conditions, medication use, their dietary analysis (by 3-days food recalls), gut microbiota and fecal metabolome. The direct (face to face) monitoring sessions will be conducted at the enrollment, one month, two months and at the end of the study (at the third month) by giving routine clinical care to all enrolled babies, which included physical examination, growth monitoring, health, and nutrition education (counseling on infant and young child feeding practices, personal hygiene, and hand washing). This monitoring session will be held by practitioner and nutritionist. Subjects will be chosen based of the inclusion & exclusion criteria. There are two research groups. The first group will be given pediatric nutrition care (PNC). In this group parents will receive nutritional advice about how many calories are needed, the type and form of food that can be given so that the baby can gain weight accordingly. In the second group, subject will receive PNC and food for special medically purposes/FSMP that will be given according to daily calorie needs which are determined based on ideal body weight (BB) according to body length. In general, FSMP will be given 3 times a day, according to the needs of each subject. Parents will be taught about preparation of FSMP e.g., dissolving and the correct amount of product (image will be attached in the appendix). FSMP will be given during the research period and will be discontinued when participant do not need it anymore.

Infants whose weight gain is below the 5th percentile of the WHO weight gain table and infants who are already mildly undernourished will be immediately given PNC + FSMP and not included in the PNC group. At the beginning of the study, parents will be asked about the type of food and milk consumed, amount and eating patterns, the incidence of illness such as fever, cough, runny nose, diarrhea, vomiting, sleep, and the general condition of the baby. Research team till measure body weight, length, head circumference and take the feces for microbiota and metabolome examination before intervention. Feces obtained will be stored at temperatures below 5ºC for a maximum of 24 hours. Subjects will be monitored for 4 weeks. In the fourth weeks there will be an examination of body weight, length, episodes of illness and stool collection for the second examination of microbiota and metabolome. At the end of the first month intervention, the investigators will ask the parents for giving permission to draw the blood from their children to see the plasma metabolome.

If within 4 weeks, the baby has gained a good weight gain according to the existing table (above P 15), then the subject does not need to take FSMP again but will continue to be monitored every month to prevent the second growth faltering event. If the baby is initially in the PNC group and does not gain good weight, PNC + FSMP will be given. The intervention and monitoring will be done for a total of 12 weeks. Every week, the total volume that had been consumed will be monitored by the field assistant by phone. Product acceptance questionnaires for the FSMP product will be assessed using a questionnaire during the monitoring visits at visit 1, 2 and 3. The occurrence of adverse events and medication use was recorded throughout the whole study period. All subjects will be provided with BPJS insurance during the study period up to one month after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* Weight faltering babies (weight increments below percentile 15th of weight increments table WHO age 6-12 month-old with good nutritional or mild undernutrition status
* Have a growth chart monitoring (weight, length and head circumference) at least one time (at birth).
* Have the data of height and weight from father and mother (genetic height potential)
* No major congenital anomaly, severely stunted at birth, not having thyroid problem, not suffered from prominent gastrointestinal diseases, severe diseases at the time of inclusion (severe pneumonia, severe dehydration, etc)
* Not suffered from parasitic manifestation by examining the faecel sample at the time of recruitment
* Parents want to follow the study by signing the informed consent

Exclusion Criteria:

* Subjects with stunting
* Subject in the severe disease condition at the time of recruitment
* Severe acute malnutrition
* Parents do not want to participate in the study
* Presence of cow's milk allergy
* Presence of lactose intolerance
* Presence of galactosemia
* Condition needing a special diet, like major renal and hepatic dysfunction
* Have conditions that will influence the nutritional status such as moderate to severe dehydration, organomegaly, oedema.
* Babies with weight more than ideal body weight

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 188 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Weight increment difference in grams | one month
  to look for the relative efficacy of PNC and PNC + FSMP (SGM 100) on the weight increments

SECONDARY OUTCOMES:
weight increment percentile | during study period (3 months)
  to look for the improvement of weight increments percentile of all subjects measured from time to time during the study period
length increments in cm | during study period (3 months)
  to look length increments of all subjects measured from time to time during the study period
body mass index in kg/m^2 | during study period (3 months)
  to look length increments and body mass index alteration of all subjects measured from time to time during the study period
Composition (proportion) of each type of microorganisms in fecal | baseline, one month
  changes of fecal microbiome composition (proportion of microorganisms' type) in control and intervention group
level of metabolites in faecal (faecal metabolome) | baseline and one month in the study
  level of metabolites in untargetted faecal metabolome analysis measured by LCMS in control and intervention group
Number of children with existence of any medical health history to understand any related risk factors of weight faltering (obtained from anamnesis and physical examination) | at screening, baseline, one month, second month and third month
  identify medical health history (obtained from anamnesis and physical examination) to understand any related risk factors of weight faltering during study period and from health history starting from prenatal, including their delivery mode, gestational age
Amount of Energy intake of children | at baseline, one month, and second month of the study
  quantifying amount of energy intake among children in the study measured by dietary recall using interview
Number of children who accept the product | during study period (at one month, second month and third month)
  acceptance of the product during study period measured by the proportion of respondents who answer all questions in acceptance questionnaire with agree or strongly agree
Number of children who tolerate the product | during study period (at one month, second month and third month)
  tolerance of the product during study period measured by the proportion of children who were consuming the recommended amount of product during the study without any adverse event related to the consumption
compliance of the product consumption | during study period (at one month, second month and third month)
  compliance of the product consumption during study period measured by the proportion of children who were consuming the recommended amount of product during the study
infection episodes | during study period (at one month, second month and third month)
  number of infection incidence experienced by children during study period
sleep quality | during study period (at one month, second month and third month)
  the mean duration of sleep of children during study period recorded by a diary during study period (by calculating the mean duration of the sleep)

CONTACTS AND LOCATIONS:
Overall Officials: Conny Tanjung, MD, PhD, Principal Investigator — Hasanuddin University
Locations (1):
- Hasanuddin University, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No